CLINICAL TRIAL: NCT01045057
Title: Clinical Feasibility of a New Surgical Tool for Primary or Secondary Tracheoesophageal Puncture and Voice Prosthesis Insertion for Prosthetic Voice Rehabilitation After Total Laryngectomy
Brief Title: Clinical Feasibility of New Tracheoesophageal Puncture Set
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Atos Medical AB (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UD743_FRITZ_MULTI
Record Dates: First submitted 2010-01-06; First posted 2010-01-08 (Estimated); Results first posted 2015-02-10 (Estimated); Last update posted 2021-06-11 (Actual); Status verified 2021-06

CONDITIONS: Larynx Cancer
Keywords: voice prosthesis, larynx cancer, laryngectomy
MeSH Terms: conditions — Laryngeal Neoplasms

STUDY DESIGN:
Intervention Model Description: Provox Vega Puncture Set
Oversight: Data Monitoring Committee: No

ARMS (1):
- Puncture Set and Flexible Protector (Experimental): Provox Vega Puncture Set is used to create the primary puncture and insert the prosthesis during total laryngectomy
  Interventions: Device: Puncture Set and Flexible Protector

INTERVENTIONS:
Device: Puncture Set and Flexible Protector — The Provox Vega Puncture Set will be used to create the tracheoesophageal puncture and place the voice prosthesis. In secondary punctures the Provox Flexible Protector may be used for pharynx protection.

SUMMARY:
During a total laryngectomy a puncture is created in the tracheoesophageal wall and a voice prosthesis is inserted. With this voice prosthesis the patient learns to speak again. During this study a new surgical tool will be investigated that creates the puncture and places the voice prosthesis.

ELIGIBILITY:
Inclusion Criteria:

* primary puncture during total laryngectomy
* secondary puncture some time after total laryngectomy

Exclusion Criteria:

* anatomical abnormalities that prevent appropriate pharynx protection during secondary puncture
* not eligible to use a voice prosthesis for other reasons

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2009-12; Primary Completion 2011-03 (Actual); Study Completion 2011-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Frans JM Hilgers, MD, PhD, Principal Investigator — The Netherlands Cancer Institute
Locations (5):
- University Hospital Leuven, Leuven, Belgium
- Bundeswehr Krankenhaus, Ulm, Germany
- Netherlands (2):
  - Netherlands Cancer Institute, Amsterdam, North Holland
  - Erasmus Medical Center, Rotterdam, South Holland
- Hospital de la Santa Creu I Sant Pau Universitat Autònoma de Barcelona, Barcelona, Spain

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Prospective study, carried out in 5 different medical centers in 4 different countries. Recruitment period runs from November 2009-March 2011
Groups:
- Provox Vega Puncture Set: Patients with laryngeal cancer and a total laryngectomy in whom a puncture was made and a voice prosthesis was placed by means of the Provox Vega Puncture Set
Period: Overall Study
Arm/Group | Provox Vega Puncture Set
Started | 27
Completed | 27
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- Provox Vega Puncture Set: Group of larynx cancer patients undergoing a total laryngectomy whereby the puncture and placement of the voice prosthesis is done with the Provox Vega Puncture Set
Arm/Group | Provox Vega Puncture Set
Number analyzed (Participants) | 27
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 18
  >=65 years | 9
Age, Continuous [Mean (Standard Deviation); unit: years] | 62 (7.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 23
Region of Enrollment [Number; unit: participants]
  Spain | 2
  Belgium | 7
  Germany | 13
  Netherlands | 5

OUTCOME MEASURES:

1. Primary Outcome: Success Rate of Procedure
Description: As successful counted all successful procedures in which the tracheal flange of the voice prosthesis unfolded completely without help of additional tools. A success rate of 80% and higher was considered acceptable.
Time Frame: immediate observation during surgery
Population: Number subjects based on optimal minimax two-stage design. Based on power calculation, 26 patients should be included. In first stage, 20/23 successful insertions are needed to continue. In second stage, with 23/26 successful insertions device is considered safe. Analysis is per protocol.
Measure: Number; unit: Nr part. with succesful insertions
Groups:
- Provox Vega Puncture Set: Patients with laryngeal cancer and a total laryngectomy in whom a TE puncture was made and a voice prosthesis was placed by means of the Provox Vega Puncture Set
Arm/Group | Provox Vega Puncture Set
Number analyzed (Participants) | 27
Nr part. with succesful insertions | 23

2. Secondary Outcome: Satisfaction of Physician
Description: Satisfaction of the physicians with the new tools was investigated by asking them which tool set they prefer: the new set from the study or the set they would have normally used.
Time Frame: 1 month
Population: as for outcome 1
Measure: Number; unit: Number of times new set was preferred
Groups:
- Provox Vega Puncture Set: Patients in whom a voice prosthesis was placed by means of the Provox Vega Puncture Set
Arm/Group | Provox Vega Puncture Set
Number analyzed (Participants) | 27
Number of times new set was preferred | 26

3. Secondary Outcome: Cost Effectiveness Calculation
Description: cost effectiveness of the new tool set is compared to that of the set that would have been used in the absence of the new puncture set.
  Measurements are: time needed to perform procedure
Time Frame: 1 month
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | Provox Vega Puncture Set
Number analyzed (Participants) | 27
seconds | 155.4 (115.6)

4. Secondary Outcome: Postoperative Results
Description: Patients were followed-up one month after surgery.Patients with secondary punctures filled out a questionnaire.
Time Frame: 1 month
Population: Only patients with secondary puncture filled out questionnaire. Seven patients had secondary puncture. One patient refused to fill out questionnaire. Six patients remained. Analysis per protocol.
Measure: Number; unit: Number of patients
Groups:
- Secondary Puncture: Patients who had a secondary puncture
Arm/Group | Secondary Puncture
Number analyzed (Participants) | 6
Number of patients
  Satisfisfied with procedure | 6
  Would recommend procedure | 6

ADVERSE EVENTS:
Time Frame: During one month after the surgery
Description: all adverse events, including expected/non-related events were recorded
Groups:
- Provox Vega Puncture Set: Group of larynx cancer patients undergoing laryngectomy whereby the puncture and the placement of the voice prosthesis is done with the Provox Vega Puncture set
Arm/Group | Provox Vega Puncture Set
Serious Adverse Events (participants affected / at risk) | 0/27
Other Adverse Events (participants affected / at risk) | 8/27
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Provox Vega Puncture Set (N=27)
Pharyngocutaneous Fistula (Surgical and medical procedures) | 3 (3) — In all 3 patients known significant risk factors were present that are deemed to have caused the fistula. As such, these complications are not considered related to device/procedure. Fistula occurrence rate was within previously reported ranges.
Damage posterior pharyngeal wall (Surgical and medical procedures) | 1 (1) — Posterior pharyngeal wall was damaged during dilatation before the puncture took place. Non-device related.
Damage posterior esophageal wall (Surgical and medical procedures) | 1 (1) — Puncture penetrated posterior esophageal wall because window of device used for pharynx protection (not part of subject device)could not be located by palpation or visualization. Event did not cause any harm to patient. Event is not device related.
Retracted voice prosthesis (Surgical and medical procedures) | 1 (1) — Voice prosthesis retracted while cleaning it, and was repositioned. No patient harm. Event is related to patient anatomy, not related to device/procedure.Occurred in home situation, can occur when voice prosthesis (e.g. due to edema) fits too tight.
Tracheitis (Surgical and medical procedures) | 1 (1) — Patient developed tracheitis, caused by COPD and the related use of Prednisone and inhalation medications. Patient received antibiotics and was fine. Event was unrelated to device.
Wound dehiscence (Surgical and medical procedures) | 1 (1) — Wound healing problems considered to be caused by pre-existing risk factors (Radiotherapy,prednisone use)and surgical risk factor of bilateral neck dissection.Not device related.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No